CLINICAL TRIAL: NCT03953235
Title: A Phase 1/2 Study of GRT-C903/GRT-R904, a Vaccine Targeting Shared Neoantigens, in Combination With Immune Checkpoint Blockade for Patients With Advanced Solid Tumors
Brief Title: A Study of a Personalized Cancer Vaccine Targeting Shared Neoantigens
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gritstone bio, Inc. (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GO-005
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Non-Small Cell Lung Cancer; Colorectal Cancer; Pancreatic Cancer; Solid Tumor; Shared Neoantigen-Positive Solid Tumors
Keywords: neoantigen cancer vaccine; shared neoantigen; GRT-C903; GRT-R904; immunotherapy; PD-1; CTLA-4; nivolumab; ipilimumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Pancreatic Neoplasms; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1 (Experimental): * GRT-C903
  * GRT-R904
  * nivolumab
  * ipilimumab
  Interventions: Biological: GRT-C903; Biological: GRT-R904; Biological: nivolumab; Biological: ipilimumab
- Phase 2 (Experimental): * GRT-C903
  * GRT-R904
  * nivolumab
  * ipilimumab
  Phase 2 for some patients includes a monthly or every two month treatment schedule
  Interventions: Biological: GRT-C903; Biological: GRT-R904; Biological: nivolumab; Biological: ipilimumab

INTERVENTIONS:
Biological: GRT-C903 — a shared neoantigen cancer vaccine prime
Biological: GRT-R904 — a shared neoantigen cancer vaccine boost
Biological: nivolumab — anti-PD-1 monoclonal antibody
Biological: ipilimumab — anti-CTLA-4 monoclonal antibody

SUMMARY:
The purpose of this study is to evaluate the dose, safety, immunogenicity and early clinical activity of GRT-C903 and GRT-R904, a neoantigen-based therapeutic cancer vaccine, in combination with immune checkpoint blockade, in patients with advanced or metastatic non-small cell lung cancer, microsatellite stable colorectal cancer, pancreatic cancer, and shared neoantigen-positive tumors. Based on the Phase 1 data, an updated vaccine candidate (SLATE-KRAS or version 2) was developed that removed 16 of the 20 mutations included in the original vaccine (version 1) and solely targets KRAS mutations.

DETAILED DESCRIPTION:
Tumors harboring non-synonymous deoxyribonucleic acid (DNA) mutations can present peptides containing these mutations as non-self antigens in the context of HLA on the tumor cell surface. A fraction of mutated peptides result in neoantigens capable of generating T-cell responses that exclusively target tumor cells. Some of these tumor-specific neoantigens are known or expected to be common across a subset of patients and are called shared neoantigens. This study aims to target shared neoantigens using a heterologous prime/boost therapeutic vaccine approach (GRT-C903 first followed by GRT-R904) in combination with checkpoint blockade to stimulate an immune response. This study will explore the safety and early clinical activity of this neoantigen-based immunotherapy intended to induce T-cell responses specific for the shared neoantigens contained within the therapeutic vaccine. Phase 1 will test multiple doses and combinations with checkpoint blockade and Phase 2 will test for early signs of clinical activity using a vaccine regimen based on Phase 1 data.

ELIGIBILITY:
Inclusion Criteria:

* Provide a signed and dated informed consent form prior to initiation of study-specific procedures.
* Patients with the indicated advanced or metastatic solid tumor as follows:

  1. Microsatellite-stable colorectal cancer (MSS-CRC) who are currently receiving systemic treatment with a fluoropyrimidine and oxaliplatin and/or irinotecan that may include a VEGF or EGFR targeting therapy as their 1L therapy for metastatic disease OR who have experienced disease progression following treatment with a fluoropyrimidine, oxaliplatin, and irinotecan that may include a VEGF or EGFR targeting therapy and have not received additional lines of systemic therapy in the metastatic setting.
  2. Non-small cell lung cancer (NSCLC) who are currently receiving systemic treatment with an anti-PD-(L)1 antibody in combination with cytotoxic, platinum-based chemotherapy OR who have experienced disease progression following treatment with an anti-PD-(L)1 antibody in combination with cytotoxic, platinum-based chemotherapy (or anti-PD-(L)1 alone if patient refuses platinum-based chemotherapy), and have not received additional lines of systemic therapy in the metastatic setting.
  3. Pancreatic ductal adenocarcinoma (PDA) who are currently receiving systemic cytotoxic chemotherapy as their 1L therapy for metastatic disease OR who have experienced disease progression on 1L systemic cytotoxic chemotherapy and have received no more than 1 prior line of therapy in the metastatic setting.
  4. Any solid tumor histology where the patient has experienced disease progression with all available therapies known to confer clinical benefit
* Patient's tumor possesses one of the mutations listed below, and is determined to express a HLA allele for antigen presentation of the identified tumor mutation:

VERSION 1.0 of the expression cassette:

BRAF_G466V // CTNNB1_S37F // CTNNB1_S45F // CTNNB1_S45P // CTNNB1_T41A // ERBB2_Y772_A775dup // KRAS_G12C or NRAS_G12C // KRAS_G12D or NRAS_G12D // KRAS_G12V // KRAS_G13D // KRAS_Q61H or NRAS_Q61H // KRAS_Q61K or NRAS_Q61K // KRAS_Q61L or NRAS_Q61L // KRAS_Q61R or NRAS_Q61R // TP53_K132E // TP53_K132N // TP53_R213L // TP53_R249M // TP53_S127Y

VERSION 2.0 of the expression cassette:

KRAS_G12C or NRAS_G12C // KRAS_G12D or NRAS_G12D // KRAS_G12V or NRAS_G12V // KRAS_Q61H or NRAS_Q61H

* ECOG Performance Status 0 or 1
* Measurable disease according to RECIST v1.1
* Adequate organ function, as measured by laboratory values (criteria listed in protocol)

Exclusion Criteria:

* Tumors with genetic characteristics as follows:

  1. For NSCLC, patients with a known genetic driver alteration in EGFR, ALK, ROS1, RET, or TRK
  2. Patients with known MSI-high disease based on institutional standard
* Known exposure to chimpanzee adenovirus or any history of anaphylaxis in reaction to a vaccination
* Bleeding disorder (eg., factor deficiency, coagulopathy) or history of significant bruising or bleeding following IM injections or blood draws
* History of allogenic/solid organ transplant
* Active, known, or suspected autoimmune disease
* Active tuberculosis or recent (<2 week) clinically significant infection, or evidence of active hepatitis B or hepatitis C
* Known history of positive test for human immunodeficiency (HIV) or known acquired immunodeficiency syndrome (AIDS)

Complete inclusion and exclusion criteria are listed in the clinical study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs), serious adverse events (SAEs), and dose limiting toxicities (DLTs) | Initiation of study treatment through 100 days post-last dose (up to approximately 27 months)
Objective Response Rate (ORR) in Phase 2 using RECIST v1.1 | Initiation of study treatment until disease progression (up to approximately 27 months)
Identify the recommended Phase 2 dose (RP2D) of GRT-C903 and GRT-R904 | Up to approximately 6 months

SECONDARY OUTCOMES:
Measure the immune response to the neoantigens encoded by GRT-C903 and GRT-R904 | Baseline to end of treatment (up to approximately 12 months)
Objective Response Rate (ORR) in Phase 1 using RECIST v1.1 | Initiation of study treatment until disease progression (up to approximately 27 months)
Duration of response (DOR) using RECIST v1.1 | Initiation of study treatment until disease progression (up to approximately 27 months)
Clinical benefit rate (CBR) using RECIST v1.1 | Initiation of study treatment until disease progression (up to approximately 27 months)
Progression-free survival (PFS) | Up to approximately 4 years
Overall survival (OS) | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - UCLA Medical Center, Santa Monica, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Chicago Medicine, Comprehensive Cancer Center, Chicago, Illinois
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Columbia University Medical Center, Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia

REFERENCES:
- [Derived] Rappaport AR, Kyi C, Lane M, Hart MG, Johnson ML, Henick BS, Liao CY, Mahipal A, Shergill A, Spira AI, Goldman JW, Scallan CD, Schenk D, Palmer CD, Davis MJ, Kounlavouth S, Kemp L, Yang A, Li YJ, Likes M, Shen A, Boucher GR, Egorova M, Veres RL, Espinosa JA, Jaroslavsky JR, Kraemer Tardif LD, Acrebuche L, Puccia C, Sousa L, Zhou R, Bae K, Hecht JR, Carbone DP, Johnson B, Allen A, Ferguson AR, Jooss K. A shared neoantigen vaccine combined with immune checkpoint blockade for advanced metastatic solid tumors: phase 1 trial interim results. Nat Med. 2024 Apr;30(4):1013-1022. doi: 10.1038/s41591-024-02851-9. Epub 2024 Mar 27. PMID 38538867